CLINICAL TRIAL: NCT07335224
Title: MPOWER: A Pilot Trial Among Men With Prostate Cancer: Optimizing Wellness by Enhanced Relief From Hot Flashes With Acupuncture
Brief Title: Men With Prostate Cancer: Optimizing Wellness by Enhanced Relief From Hot Flashes With Acupuncture
Acronym: MPOWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INOVA-2025-152
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Hot Flashes; Acupuncture Therapy; Vasomotor Symptoms; Androgen Deprivation Therapy; Prostatic Neoplasms
MeSH Terms: conditions — Hot Flashes; Prostatic Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: A total of 24 men with prostate cancer receiving ADT will be randomly assigned to one of two groups: one group will begin acupuncture right away, and the other group will begin acupuncture after a delay, with regular check-ins during the waiting period. All participants will receive standard lifestyle education.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Start Acupuncture (Experimental): Participants randomized to the immediate start acupuncture (IA) arm will receive a 10-week standard acupuncture protocol, consisting of weekly 30-minute sessions, in addition to lifestyle education per usual care. Acupuncture will be delivered by a certified acupuncturist with expertise in oncology care. Following completion of the 10-week acupuncture period, participants will enter a 12-week follow-up phase during which no acupuncture treatments will be provided.
  Interventions: Other: Acupuncture
- Delayed Start Acupuncture (Active Comparator): Participants randomized to the delayed start acupuncture (DA) arm will receive lifestyle education per usual care without acupuncture during the initial 10-week comparison period. Beginning at week 12, participants will initiate the same 10-week standard acupuncture protocol, consisting of weekly 30-minute sessions delivered by a certified acupuncturist with expertise in oncology care.
  Interventions: Behavioral: Lifestyle Management

INTERVENTIONS:
Other: Acupuncture — Acupuncture is a form of alternative medicine and a component of traditional Chinese medicine (TCM) in which thin needles are inserted into the body
  Arms: Immediate Start Acupuncture
Behavioral: Lifestyle Management — lifestyle education per usual care without acupuncture for the first 10 weeks. At week 12, they will begin the acupuncture protocol (weekly 30-minute sessions).
  Arms: Delayed Start Acupuncture

SUMMARY:
Prostate cancer is the most common cancer among men in the United States. Many men with prostate cancer are treated with hormone therapy, also called androgen deprivation therapy (ADT). While this treatment is effective, it often causes bothersome side effects such as hot flashes, poor sleep, fatigue, and other physical and emotional symptoms. There is currently no standard treatment to help manage these side effects in men. Acupuncture is a non-drug treatment that has been shown to help reduce hot flashes and related symptoms in women receiving hormone therapy for breast cancer. However, much less is known about whether acupuncture is helpful for men receiving hormone therapy for prostate cancer. This study will test whether an acupuncture program, combined with usual lifestyle education, is feasible and acceptable for men undergoing ADT. The study will also explore whether acupuncture may help reduce hot flashes and improve related symptoms. A total of 24 men with prostate cancer receiving ADT will be randomly assigned to one of two groups: one group will begin acupuncture right away, and the other group will begin acupuncture after a delay, with regular check-ins during the waiting period. All participants will receive standard lifestyle education. Participants will be followed for about five months and will be asked to complete daily hot flash diaries, questionnaires about their symptoms and quality of life, and wear a Fitbit to track sleep. The results of this pilot study will help determine whether a larger study should be conducted to better understand the role of acupuncture in managing hormone therapy side effects in men with prostate cancer.

DETAILED DESCRIPTION:
This study is a pilot feasibility randomized controlled trial designed to evaluate the acceptability, feasibility, and delivery of an acupuncture intervention for men with prostate cancer receiving androgen deprivation therapy (ADT). A total of 24 participants will be enrolled and randomized in a 1:1 ratio to either an intervention arm with immediate acupuncture (IA) or a wait-list attention control arm with delayed acupuncture (DA), resulting in 12 participants per group. Randomization will be conducted using a simple randomization scheme.

Participants will be followed for a total of 22 weeks. Those assigned to the IA arm will receive a standardized acupuncture protocol consisting of weekly 30-minute manual acupuncture sessions for 10 weeks, administered by a certified acupuncturist with expertise in oncology care. In addition to acupuncture, participants in the IA arm will receive lifestyle education consistent with usual clinical practice. Following completion of the 10-week acupuncture period, participants in the IA arm will enter a 12-week follow-up phase without acupuncture treatment.

Participants assigned to the DA arm will receive lifestyle education per usual care during the initial 10-week period without acupuncture, along with scheduled check-ins with study staff to control for attention. At week 12, participants in the DA arm will begin the same standardized acupuncture protocol as the IA arm, consisting of weekly 30-minute sessions for 10 weeks. This design allows all participants to receive the acupuncture intervention while enabling comparison of feasibility and acceptability between immediate and delayed initiation.

ELIGIBILITY:
Inclusion Criteria:

* Male
* At least 18 years of age
* Histologically or cytologically confirmed adenocarcinoma of prostate of any stage I-IV
* Undergoing androgen deprivation therapy (ADT) and/or androgen receptor pathway inhibitors
* Experiencing moderate to severe daily interference from hot flashes, as indicated by the Hot Flash Related Daily Interference Scale (score≥4)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Able to read, understand, and provide written informed consent

Exclusion Criteria:

* Severe or uncontrolled concurrent disease, infection or co-morbidity that, in the opinion of the Investigator, would make the patient inappropriate for enrollment
* Known hypersensitivity to the acupuncture needles
* Any condition that in the opinion of the Investigator would impair the patients' ability to comply with the study procedures
* Unable to comply with study requirements
* Use of acupuncture for hot flashes within 6 months prior to enrollment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Study feasibility - patient enrollment | 12 months
  Study feasibility will be measured by patient enrollment rates, defined as the proportion of eligible patients approached about the study who consent to participate.
Study feasibility - Patient intervention engagement | 18 months
  Study feasibility will be measured by patient intervention engagement, defined as the proportion of enrolled patient subjects who attend at least 6 of 10 scheduled acupuncture visits.

SECONDARY OUTCOMES:
Intervention acceptability - quantitative | 11, 17, and 22 weeks
  Intervention acceptability will be measured using satisfaction ratings.
Intervention acceptability - qualitative | 22 weeks
  Intervention acceptability will be evaluated using thematic analysis of post-intervention semi-structured interviews.
Hot Flash Severity Score | Baseline, 11, 17, and 22 weeks
  The primary patient outcome is the weekly mean hot flash score, which is calculated by multiplying hot flash frequency by severity, as recorded in the Daily Hot Flash Diary (DHFD).

CONTACTS AND LOCATIONS:
Overall Officials: Jeanny Aragon-Ching, MD, Principal Investigator — Inova Schar Cancer
Locations (1):
- Inova Schar Cancer Institute, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Data will be available upon reasonable request.